CLINICAL TRIAL: NCT01102621
Title: Hearing Loss and Complaint in Patients With Head and Neck Cancer Treated With Radiotherapy
Status: Completed | Type: Observational
Sponsor: Hospital A.C. Camargo (Other)
Responsible Party: Hearing loss and Complaint in patients with head and neck cancer treated with radiotherapy, Hospital A C Camargo
Other Study IDs: HL1
Record Dates: First submitted 2010-04-06; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-03

CONDITIONS: Hearing Loss
Keywords: hearing loss; head and neck cancer; radiotherapy; hearing complaint; Hearing loss due to the exposure of radiotherapy
MeSH Terms: conditions — Hearing Loss; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case-control, head and neck cancer with radiotherapy: The group of exposed individuals had to be patients with disease-free survival interval of at least two years subsequent to treatment for head and neck cancer by means of radiotherapy alone or in combination, in which the auditory system was included in the field of irradiation.
- case-control, head an neck cancer without radiotherapy: The group of non-exposed individuals (control group) had to be patients who had not undergone oncological treatment that put their hearing at risk and who were age-matched (2 years). This group was formed by individuals who had had pelvic tumors or skin tumors and who had only undergone local surgery to remove their tumors, and by female volunteers from the hospital. All of these individuals were asked whether they would be willing to participate in a study, without knowing in advance whether they had any previous hearing problems or complaints.

SUMMARY:
Hypothesis: Treatment for head and neck tumors often involve methods that affect the auditory system and cause hearing loss. Neck dissection negatively impacts the lymphatic drainage, chemotherapy uses ototoxic drugs, radiotherapy affects blood flow and tissue radiation is toxic to the ear and may lead to hearing losses of various types and degrees.

Objective: To investigate occurrences of hearing loss and complaints among patients with head and neck tumors who underwent radiotherapy.

Study design: Prospective, case-control study. Setting: Tertiary care center hospital.

Subjects and Methods: 282 subjects were evaluated, 141 with head and neck tumors and 141 as an age-matched control group. The controls had never undergone oncological treatment that put their hearing at risk. All subjects underwent audiological evaluation, including the HHIE questionnaire, pure tone audiometry, speech audiometry and immittance audiometry. The radiation dose received by the auditory system was calculated based on the percentage of the external auditory canal included in the radiation field.

ELIGIBILITY:
Inclusion Criteria:

* The group of exposed individuals
* had to be patients with disease-free survival interval of at least two years subsequent to treatment for head and neck cancer
* radiotherapy alone or in combination, in which the auditory system was included in the field of irradiation.
* The group of non-exposed individuals (control group)
* had to be patients who had not undergone oncological treatment that put their hearing at risk
* age-matched (2 years). This group was formed by individuals who had had pelvic tumors or skin tumors and who had only undergone local surgery to remove their tumors, and by female volunteers from the hospital.
* All of these individuals were asked whether they would be willing to participate in a study, without knowing in advance whether they had any previous hearing problems or complaints.

Exclusion Criteria:

* congenital hearing loss
* otological surgery

Ages: 11 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study design: Prospective, case-control study. Setting: Tertiary care center hospital.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The hearing loss was evaluated through conventional tone threshold audiometry and a questionaire of hearing handicap was applied to both groups (individuals exposed to radiotherapy and the control group). | patientes were evaluated two years after finished the treatement
  We observed mild to moderate hearing losses at frequencies of 57.4% in right ears and 59.6% in left ears in the group exposed to radiotherapy and in the control group, 43.3% ofmild to moderate hearing loss in both ears.Severe or profound hearing losses or anacusis occurred at frequencies of 6.4% in right ears and 8.5% in left ears, versus only 1.4% in the control group.Furthermore, severe handicap was observed in 2.8% of the individuals in the control group, versus 19.1% in the group exposed to radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital A C Camargo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Schultz C, Goffi-Gomez MV, Pecora Liberman PH, Pellizzon AC, Carvalho AL. Hearing loss and complaint in patients with head and neck cancer treated with radiotherapy. Arch Otolaryngol Head Neck Surg. 2010 Nov;136(11):1065-9. doi: 10.1001/archoto.2010.180. PMID 21079158